CLINICAL TRIAL: NCT02180841
Title: Effect of Soy on HDL-C Function, Central Blood Pressure, and Arterial Stiffness
Acronym: SOY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: PKE SOY
Record Dates: First submitted 2014-06-23; First posted 2014-07-03 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
Keywords: soy; hypertension; HDL-C; cholesterol efflux; cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Soy 25g (Experimental): Soy protein powder (25g/day)
  Interventions: Dietary Supplement: Soy Protein Powder (25g/d); Dietary Supplement: Placebo; Dietary Supplement: Soy Protein Powder (50g/d)
- Soy 50g (Experimental): Soy protein powder 50 g/day
  Interventions: Dietary Supplement: Soy Protein Powder (25g/d); Dietary Supplement: Placebo; Dietary Supplement: Soy Protein Powder (50g/d)
- Control (Placebo Comparator): Control powder
  Interventions: Dietary Supplement: Soy Protein Powder (25g/d); Dietary Supplement: Placebo; Dietary Supplement: Soy Protein Powder (50g/d)

INTERVENTIONS:
Dietary Supplement: Soy Protein Powder (25g/d) — Participants will consume 25g soy protein powder daily for a 6 week treatment period.
Dietary Supplement: Placebo — Participants will consume a placebo control powder containing 0g soy protein powder daily for a 6 week treatment period.
Dietary Supplement: Soy Protein Powder (50g/d) — Participants will consume 50g soy protein powder daily for a 6 week treatment period.

SUMMARY:
The purpose of the proposed pilot study is to evaluate the effects of a soy protein isolate with naturally occurring isoflavones on the properties of HDL-C (total HDL-C, HDL particle size and HDL function), central blood pressure, and indices of arterial stiffness.

DETAILED DESCRIPTION:
The investigators propose to conduct a randomized three-period, crossover study to evaluate the effect of soy protein supplementation on HDL function. To ensure that there are no effects of treatment order on outcome measures, subjects will be randomized to a treatment sequence. Healthy males and females (n = 20; 35 to 60 years of age) with systolic blood pressure greater than 120 mm Hg and/or diastolic blood pressure greater than 80 mm Hg will be recruited for this study. Subjects will undergo 3 treatment periods in random order. These treatment periods will include: A) 25 g/d soy protein powder; B) 50 g/d soy protein powder; C) 0 g/d protein powder (control). Each treatment will be provided for 6 weeks separated by a 2-week break between treatment periods. All subjects will be encouraged to maintain body weight and physical activity levels during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* 35-60 years old,with
* Systolic blood pressure greater than 120 mm Hg
* Diastolic blood pressure greater than 80 mm Hg
* BMI within 18-39 kg/m2 ,
* non smokers with
* no inflammatory diseases and
* not taking medication for high cholesterol, blood pressure, or glucose control

Exclusion Criteria:

* Under 35 years of age or over 60 years old
* Systolic blood pressure <120 or Diastolic blood pressure <80
* smoker
* inflammatory disease
* BMI outside of 18-39kg/m2 range
* taking medication
* refusal to discontinue any other supplement use

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
HDL function (RCT) as measured by cholesterol efflux. | Baseline
  Prior to start of intervention
HDL function (RCT) as measured by cholesterol efflux. | Week 6
  End of treatment 1
HDL function (RCT) as measured by cholesterol efflux. | Week 14
  End of treatment 2
HDL function (RCT) as measured by cholesterol efflux. | Week 22
  End of treatment 3

SECONDARY OUTCOMES:
HDL particle size | Baseline
  Prior to start of intervention
HDL particle size | Week 6
  End of treatment 1
HDL particle size | Week 14
  End of treatment 2
HDL particle size | Week 22
  End of treatment 3

OTHER OUTCOMES:
Lipids (including lipoproteins and apolipoproteins) | Baseline
  Prior to start of intervention
Lipids (including lipoproteins and apolipoproteins) | Week 6
  End of treatment 1
Lipids (including lipoproteins and apolipoproteins) | Week 14
  End of treatment 2
Lipids (including lipoproteins and apolipoproteins) | Week 22
  End of treatment 3
Central blood pressure (including augmentation index, pulse pressure, and pulse wave velocity). | Baseline
  Prior to start of intervention
Central blood pressure (including augmentation index, pulse pressure, and pulse wave velocity). | Week 6
  End of treatment 1
Central blood pressure (including augmentation index, pulse pressure, and pulse wave velocity). | Week 14
  End of treatment 2
Central blood pressure (including augmentation index, pulse pressure, and pulse wave velocity). | Week 22
  End of treatment 3

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States